CLINICAL TRIAL: NCT00459264
Title: Prevention of Mood Disorders by Folic Acid Supplementation
Acronym: PRE-EMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, ProfessorJohnGeddes, Professor of Psychiatry, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 04/Q1604/110; 04T-496; 2004-003341-40; 21584/0206/001-0001
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Depression; Bipolar Disorder
Keywords: Folic Acid; Prevention; Depression; Bipolar Disorder; Teenagers
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Folic Acid
  Interventions: Drug: Folic Acid
- 2 (Placebo Comparator): Matching placebo for folic acid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Folic Acid — Folic acid oral solution 2.5mg/5ml daily for up to 3 years
  Other Names: Lexpec PL 0427/0034
  Arms: 1
Drug: Placebo — Matching placebo for folic acid oral solution (2.5mg/5ml)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether daily folic acid supplements can prevent new episodes of mood disorder in young people (aged 14-24 years) of biological parents with current or past history of depression or bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder and recurrent major depression are life-long disabling illnesses that often first become clinically apparent in the late teenage years or early twenties. People who develop clinical mood disorders characteristically have milder, short-lived symptoms of mood disturbance prior to the onset of clinical illness. These sub-clinical disturbances represent a risk factor for the subsequent development of clinical disorders (Angst 2000; Aalto-Setala, 2002). A number of physiological abnormalities associated with depression persist after symptom resolution, suggesting that depression may cause a kind of biological "scarring" of the brain that can predispose to further episodes of illness.

Nutritional supplements are a feasible intervention for primary prevention because they are likely to be acceptable and intuitively would seem to have a greater chance of being effective at a preventative stage, rather than later when disease progression has occurred.

Folate and mood disturbance

Low plasma and red cell folate have long been associated with clinical depressive disorders and treatment with folic acid (500mcg daily) has been shown to improve the therapeutic effect of fluoxetine in depressed patients (see Coppen and Bailey, 2000). A growing number of epidemiological studies also suggest links between low folate status, increased homocysteine and depressive symptomatology in the general population (Tiemeier et al, 2002; Bjelland et al, 2003; Morris et al, 2003).

Objectives

Primary

• To determine whether folic acid supplementation can prevent new episodes of mood disorder in teenage children of parents with recurrent depression or bipolar disorder

Secondary

* To determine whether folic acid supplementation can improve depression scores on the Mood and Feeling Questionnaire in teenage children of parents with recurrent depression or bipolar disorder
* To determine whether folic acid supplementation can improve scores on the Altman Mania Rating Scale in teenage children of parents with recurrent depression or bipolar disorder
* To determine whether there is a correlation between genotypes for folate enzymes and response to folate

Endpoints

Primary

• Occurrence of an episode of Axis 1 mood disorder on DSM-IV as determined by the Structured Clinical Interview for DSM-IV (SCID)

Secondary

* Change in Score on The Mood and Feeling Questionnaire
* Change in score on the Altman Mania Rating Scale
* Correlation between genotypes for folate enzymes and response to folate

Study design

This will be a randomized, concealed allocation, placebo-controlled study with masking of participants and investigators. Participants will initially enter a 4 week run-in phase during which they take folic acid (2.5mg). If consent and compliance are maintained during the active run-in, participants with then be randomised to one of two treatments in a parallel group design (a) Folic acid (2.5mg daily) or (b) identical placebo liquid. A web-based algorithm will be used which will be accessed by researchers either online or by phone call to the study office. Access to the randomisation code will be limited to the trial programmer with temporary access given to another member of the trial team during her absence. The treatment period will be thirty six months.

PRE-EMPT will continue screening until there are 200 teenagers in the randomised phase, male and female (14-24 years of age) who have a biological parent with a life-time history of recurrent major depression, bipolar I or bipolar II disorder. Family history will be assessed using proband questions. Subjects will be excluded if they have any current or past DSM-IV Axis I disorder. This will be assessed using the Structured Clinical Interview for DSM-IV (SCID). Current or past sub-syndromal mood and anxiety disorder will not be a reason for exclusion but will be assessed and used in the minimization process.We will also exclude subjects with a significant on-going medical condition, particularly epilepsy or those who are already using folate supplements and who are unwilling to give them up for the duration of the study. All subjects will give informed written consent to the study and a parent or guardian will also give written consent where subjects are under 16 years of age. Minimization will be carried out for age, gender, family history and the presence of sub-syndromal mood disturbance to ensure balanced treatment allocation.

Ratings and follow-up On entry to the study subjects will complete ten self-rating instruments, the Mood and Feeling Questionnaire (MFQ), a 32-item scale designed to detect and monitor adolescent depression in the community (Cooper and Goodyer, 1993; Wood et al, 1995). Subjects will also complete the Altman Mania Rating Scale, a 5-item scale designed to mania (Altman et al, 1997), the Insomnia Severity Index (ISI), a 5-item scale designed to detect the severity of insomnia (Morin 1993), and the Hospital Anxiety and Depression Scale (HADS) a 14 item scale to determine anxiety and depression (Zigmond and Snaith 1983). Subsequently subjects will complete the MFQ, Altman, ISI and HADS monthly. We will have available both web-based assessments and written forms, whichever the participant prefers. The other rating scales to be completed on entry are the Cambridge Life Events Rating Scale (CLE), Eysenck Personality Questionnaire (EPQ), Response Styles Questionnaire (RSQ), Parental Bonding Inventory (PBI), Children's Attributional Style Questionnaire (CAS). and the Morningness-Eveningness Questionnaire (MEQ).

At six monthly intervals subjects will be re-interviewed with the SCID to assess whether they have met criteria for any DSM-IV Axis I disorder in the preceding six months. The CLE and CAS will also be repeated at six monthly intervals.

Prior to entry to the investigation we ask subjects to provide a blood sample for the following:

1. Full blood count, Red cell folate, B12, homocysteine levels
2. DNA sample for polymorphisms of the proteins involved in folate metabolism and related neurotransmitters.

These measures (apart from the DNA analysis) will be repeated annually.

Prior to entry we also wish to assess waking salivary cortisol. In a separate study we have found that healthy young people with a parent who has a history of mood disorder (ie the same participant population that we are recruiting for this study) have elevated waking levels of salivary cortisol relative to controls.The measurement of waking salivary cortisol is a simple non-invasive test which may represent a marker of vulnerability to depression. If this is the case it might be altered by folate treatment which we are using in the present study to decrease the risk of depression.

We therefore propose to ask subjects to take a sample of waking salivary cortisol before they begin folate/placebo treatment and again after about six months in the study. In this way we will be able to assess the effect of folate/placebo treatment on waking salivary cortisol. The eventual aim will be assess whether relative to placebo folic acid treatment lowers waking salivary cortisol and whether this is associated with decreased risk of depression.

From the point of view of storage and custody the saliva samples will be treated exactly as the blood samples taken for folate estimation.

ELIGIBILITY:
Inclusion Criteria:

* aged 14-24 years
* at least one biological parent with history of recurrent major depression or bipolar disorder
* normal blood count and serum vitamin B12 level
* provide written informed consent
* in the case of participants <16 years have a parent or guardian who will also provide written informed consent

Exclusion Criteria:

* have significant active medical illness which in the opinion of the Principal Investigator could introduce additional risk factors and/or interfere with study procedures
* have current epilepsy and/or treatment with anticonvulsant drugs
* are, or intended to become,pregnant
* have current or previous Axis 1 disorder on DSM-IV (excluding adjustment disorder)
* are currently taking folate supplements and unwilling to continue
* have known hypersensitivity to folic acid or hydroxybenzoate esters
* taking methotrexate or other drugs that affect folate function

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2005-12; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of an episode of Axis 1 mood disorder on DSM-IV as determined by the SCID | Within 3 years

SECONDARY OUTCOMES:
Change in score on the Altman Mania Rating Scale | Within 3 years
Correlation between genotypes for folate enzymes and response to folate | Baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: John R Geddes, MD FRCPsych, Principal Investigator — University of Oxford
Locations (1):
- University Department of Psychiatry, Oxford, Oxfordshire, United Kingdom